CLINICAL TRIAL: NCT01641315
Title: Immunogenicity Study of a Reduced (4-dose) Vaccine Schedule and Rabies Immunoglobulins for Post-exposure Rabies Treatment
Brief Title: Immunogenicity Study of a Reduced (4-dose) Vaccine Schedule and Rabies Immunoglobulins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal Investigator, Queen Saovabha Memorial Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC5502
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Rabies
Keywords: rabies; rabies immunoglobulin
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rabies vaccine, IM day 0,3,7,28 with RIG (Experimental): Healthy volunteers received rabies vaccination intramuscularly on day 0,3,7 and 28 with equine rabies immunoglobulin 40 IU/Kg on day 0.
  Interventions: Biological: rabies vaccine
- Rabies vaccine, IM day 0,3,7,14 with RIG (Experimental): Healthy volunteers received rabies vaccination intramuscularly on day 0,3,7 and 14 with equine rabies immunoglobulin 40 IU/Kg on day 0.
  Interventions: Biological: rabies vaccine
- Rabies vaccine, IM Day 0,3,7,14,28 with RIG (Active Comparator): Rabies exposed victims receive rabies vaccination intramuscularly on Day 0,3,7,14,28 with equine rabies immunoglobulin 40 IU/Kg on day 0
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — Group 1: rabies vaccination was given to rabies exposed victims on day 0,3,7,14,28 with ERIG on day 0.
  Group 2: rabies vaccination was given to healthy volunteers on day 0,3,7,14 with ERIG on day 0.
  Group 3: rabies vaccination was given to healthy volunteers on day 0,3,7,28 with ERIG on day 0.
  Other Names: Equine rabies immunoglobulin produced by Thai Red Cross

SUMMARY:
Reduced 4-dose intramuscular rabies vaccination schedule was announced by US-ACIP and WHO to be one of the post-exposure prophylaxis regimens. However, concurrent usage of this regimen with rabies immunoglobulin have never been studied in the aspect that the immunity level would above the protective level required by WHO (0.5 IU/ml) for at least a year period. This study would access this subject.

DETAILED DESCRIPTION:
* Controlled trial study
* All 75 volunteers who had never had rabies immunization would be enrolled and designated into 3 groups.

group 1 : 25 Healthy volunteers age 18 - 60 yr who were attacked by mammals, possible exposed to rabies and had WHO category III exposure, all receive standard post - exposure rabies treatment with 5-dose intramuscular rabies vaccine on day 0,3,7,14,28 and 40 IU/kg of equine rabies immune globulin (ERIG).

group 2 : 25 Healthy volunteers age 18 - 60 yr receive 4-dose intramuscular rabies vaccine on day 0,3,7,14 and 40 IU/kg of equine rabies immune globulin (ERIG).

group 3 : 25 Healthy volunteers age 18 - 60 yr receive 4-dose intramuscular rabies vaccine on day 0,3,7,28 and 40 IU/kg of equine rabies immune globulin (ERIG).

5 cc - Blood would be drawn from all volunteers before vaccination and on day 14, 28, 90 and 360 for rabies neutralizing antibody titers (RNab).

The GMTs of RNab among both groups would be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers age 18-60 years.

Exclusion Criteria:

* received prior rabies immunization
* pregnancy
* immunocompromised conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Rabies Neutralizing antibody titers in volunteers who receive rabies vaccination on day 0,3,7,14 | Change from baseline of Rabies Neutralizing Antibody Titers at 1 year period
  Rabies Neutralizing antibody titers in volunteers who receive rabies vaccination on day 0,3,7,14 would be determined on day 0,14, 28, 90 and 360. Rnab titers above 0.5 IU/ml would be considered as protective levels as WHO recommendation.

SECONDARY OUTCOMES:
Rabies Neutralizing antibody titers in volunteers who receive rabies vaccination on day 0,3,7,28 | Change from baseline of Rabies Neutralizing Antibody Titers at 1 year period
  Rabies Neutralizing antibody titers in volunteers who receive rabies vaccination on day 0,3,7 and 28 would be determined on day 0,14, 28, 90 and 360. Rnab titers above 0.5 IU/ml would be considered as protective levels as WHO recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Thailand